CLINICAL TRIAL: NCT02995408
Title: Development of a Resiliency Training Program for Parents of Children With Autism Spectrum Disorder
Acronym: ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Karen Kuhlthau, Associate Professor of Pediatrics, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016P002037
Record Dates: First submitted 2016-12-14; First posted 2016-12-16 (Estimated); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Stress
Keywords: resiliency training; parenting; Autism Spectrum Disorders
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental: 3RP treatment (Experimental): An adapted version of the Relaxation Response Resiliency Program (3RP) for parents of children with ASD. The adapted program incorporates the three prongs of the 3RP: RR elicitation, stress awareness, and adaptive strategies.
  Experimental arm participated in the 8-week 3RP program starting immediately after enrollment.
  Interventions: Behavioral: Relaxation Response Resiliency Program for Parents of Children with ASD
- Waitlist control (Active Comparator): An adapted version of the Relaxation Response Resiliency Program (3RP) for parents of children with ASD. The adapted program incorporates the three prongs of the 3RP: RR elicitation, stress awareness, and adaptive strategies.
  The waitlist arm participated in the 8-week 3RP program starting 3 months after enrollment.
  Interventions: Behavioral: Relaxation Response Resiliency Program for Parents of Children with ASD

INTERVENTIONS:
Behavioral: Relaxation Response Resiliency Program for Parents of Children with ASD

SUMMARY:
This study has three aims:

Phase I: Through focus group interviews with expert clinicians, leaders of organizations, and parents with children with ASD, this study aims to identify the psychosocial needs of parents of children with ASD, specifically a) the types of concerns that parents find most difficult and stressful b) areas of concern that lack support and resources, and c) areas of need for education and skill training. This study also aims to gather feedback on the Benson-Henry Institute's Relaxation Response Resiliency Program (3RP).

Phase II: Informed by Phase I findings, this study aims to develop and determine the feasibility and acceptability of a virtual 8-session Relaxation Response Resiliency (3RP) program for parents of children with ASD.

Phase II: This study also aims to test the effectiveness of a pilot wait-list control trial, establishing efficacy of a virtual resiliency program.

DETAILED DESCRIPTION:
According to the Center for Disease Control in 2012, 14.6 per 1,000 children aged 8 years old have a diagnosis of Autism Spectrum Disorder (ASD). Having a child with ASD is associated with medical expenditures of 4.1-4.6 times more than having a child without autism, and associated with 8.4-9.5 times greater general expenditures. Furthermore, children with ASD are more likely to use out-of-school behavioral health services than children without developmental or psychiatric diagnoses. Parents of children with ASD consistently show high levels of perceived distress and anxiety related to child-parent relationships, intellectual functioning, adaptive behaviors, in addition to poorer health than parents of children of typical development. These parents also exhibit significant stress related to the emotional and financial challenges of putting together treatment and future-related plans for their children. Recent studies have found a positive relationship between caregivers' stress levels while raising a child with ASD and child behavioral and conduct problems.

There is growing literature on the increased levels of parental stress associated with caring for children with ASD. One study found that caregivers of children with ASD with behavioral, hyperactivity, and emotional problems displayed atypical cortisol patterns, a biological marker of increased stress. A review article provides a comprehensive overview of the links between high levels of parental stress among parents of children with intellectual and developmental disabilities and child health and well-being. In addition to social phobias associated with children with ASD, one study even found that caring for a child with ASD showed higher stress levels for the parents correlated with the child's social impairment severity. Finally, recent studies have also found that many parents of children with ASD exhibit psychological and physical depressive symptoms. Therefore, having a children with ASD is associated with an increased risk of problems with emotional and physical health and social well-being. Resiliency is a multidimensional construct that refers to the ability to maintain adaptation and effective functioning when faced with stressors.

Resiliency provides a framework for understanding the adjustment to stress as a dynamic process. Allostasis refers to the capacity to maintain stability of physiological systems in the face of adversity. When exposed to chronic stressors, such as care for a child with ASD, individuals expend a great deal of energy attempting to maintain allostasis; this can lead to the metabolic wear and tear described as allostatic load. Evidence is accumulating that this wear and tear is mediated by changes in basal stress system activity and by effects of these changes on dependent systems. Allostatic load and resilience can therefore be assessed by measuring basal stress system activity (HPA axis and salivary alpha-amylase).

Thus, research to reduce these parents' exposure to stress and, moreover, improve parental responses to stress, may improve the wellbeing of both parents and their children. Yet, a treatment focused on the psychosocial needs in relation to stress and allostatic load of parents of children with ASD has not been developed. Research is warranted to examine and intervene upon parental stress. This study aims to design and develop a resiliency intervention to provide support to parents of children with ASD.

This intervention will be a modified version of Dr. Park's evidence-based 8-week multimodal treatment which is designed to promote adaptation to stress and promotion of resiliency. The program is an 8 session, 1-1.5 hours a week multi modal intervention that incorporates relaxation techniques, stress awareness discussion, and adaptive strategies for coping with stress. This study will refine an 8-session group virtual-delivered resiliency treatment program consisting of 8 virtual group 1-1.5 hour sessions. The goal of this study would be to advance our ultimate objective to implement a national parental resiliency program.

ELIGIBILITY:
Inclusion Criteria:

1. Being the parent of at least one child with a diagnosed autism spectrum disorder
2. Age 18 or older

Exclusion Criteria:

1. Unable or unwilling to sign the informed consent documents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-12; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuhlthau KA, Luberto CM, Traeger L, Millstein RA, Perez GK, Lindly OJ, Chad-Friedman E, Proszynski J, Park ER. A Virtual Resiliency Intervention for Parents of Children with Autism: A Randomized Pilot Trial. J Autism Dev Disord. 2020 Jul;50(7):2513-2526. doi: 10.1007/s10803-019-03976-4. PMID 30900195

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: 3RP Treatment: An adapted version of the Relaxation Response Resiliency Program (3RP) for parents of children with ASD. The adapted program incorporates the three prongs of the 3RP: RR elicitation, stress awareness, and adaptive strategies.
  Relaxation Response Resiliency Program for Parents of Children with ASD
  Experimental arm participated in the 8-week 3RP program starting immediately after enrollment.
- Waitlist Control: An adapted version of the Relaxation Response Resiliency Program (3RP) for parents of children with ASD. The adapted program incorporates the three prongs of the 3RP: RR elicitation, stress awareness, and adaptive strategies.
  Relaxation Response Resiliency Program for Parents of Children with ASD
  The waitlist arm participated in the 8-week 3RP program starting 3 months after enrollment.
Period: Overall Study
Arm/Group | Experimental: 3RP Treatment | Waitlist Control
Started | 32 | 32
Completed | 20 | 22
Not Completed | 12 | 10

BASELINE CHARACTERISTICS:
Population: Note 13 individuals were randomized but never completed the baseline survey or any intervention. (7 immediate and 6 waitlist)
Groups:
- Experimental: 3RP Treatment; Waitlist Control: An adapted version of the Relaxation Response Resiliency Program (3RP) for parents of children with ASD. The adapted program incorporates the three prongs of the 3RP: RR elicitation, stress awareness, and adaptive strategies.
  Relaxation Response Resiliency Program for Parents of Children with ASD
- Total: Total of all reporting groups
Arm/Group | Experimental: 3RP Treatment | Waitlist Control | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (7.2) | 45 (8.1) | 45 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 49
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 24 | 25 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 2 | 3
  White | 24 | 19 | 43
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 26 | 51

OUTCOME MEASURES:

1. Primary Outcome: Distress
Description: Visual Analogue Scale-Distress is a 1-item scale which asks responders to rate their level of distress on a scale of 0 to 10. A higher score indicates more distress.
Time Frame: change between baseline (week 0) to post intervention (week 12)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: 3RP Treatment | Waitlist Control
Number analyzed (Participants) | 20 | 22
score on a scale | -1.35 (2.5) | -.36 (2.74)
Statistical Analysis 1: Comparison: Experimental: 3RP Treatment vs Waitlist Control; Test type: Superiority; p = .23, t-test, 2 sided — p-value was calculated; Mean Difference (Final Values) = -.99, 95% CI 2-sided [-2.63 to 0.65]

2. Primary Outcome: Resiliency
Description: Current Experiences Scale is a 25-item measure of resilience adapted from the Post-Traumatic Growth Inventory to reflect current functioning in the domains of appreciation for life, adaptive perspectives, personal strength, spiritual connectedness, relating to others, and an additional four items to assess current adaptive health behaviors. Total scores range from 0-25 and higher scores indicate greater resilience.
Time Frame: change between baseline (week 0) to post intervention (week 12)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: 3RP Treatment | Waitlist Control
Number analyzed (Participants) | 20 | 22
score on a scale | 6.05 (8.04) | .27 (8.04)
Statistical Analysis 1: Comparison: Experimental: 3RP Treatment vs Waitlist Control; We examined between group (3RP treatment versus wait-list) differences in pre-post change scores of resiliency; Test type: Superiority; p = 0.024, t-test, 2 sided — .05 is the threshold for significance; Mean Difference (Final Values) = 5.78, 95% CI 2-sided [.78 to 10.78]

3. Primary Outcome: Stress Reactivity/Coping
Description: Measure of Current Status (MOCS-A) is a 13-item self-report measure developed to assess perceived status on ability to relax at will, recognize stress-inducing situations, restructure maladaptive thoughts, be assertive about needs, and choose appropriate coping responses. Total score range is 0 to 52, and higher scores indicate greater perceived proficiency with these skills.
Time Frame: change between baseline (week 0) to post-intervention (week 12)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Experimental: 3RP Treatment: An adapted version of the Relaxation Response Resiliency Program (3RP) for parents of children with ASD. The adapted program incorporates the three prongs of the 3RP: RR elicitation, stress awareness, and adaptive strategies.
- Waitlist Control: Waitlist for participation in an adapted version of the Relaxation Response Resiliency Program (3RP) for parents of children with ASD. The adapted program incorporates the three prongs of the 3RP: RR elicitation, stress awareness, and adaptive strategies.
Arm/Group | Experimental: 3RP Treatment | Waitlist Control
Number analyzed (Participants) | 20 | 22
score on a scale | 7.60 (7.24) | -.18 (6.66)
Statistical Analysis 1: Comparison: Experimental: 3RP Treatment vs Waitlist Control; Test type: Superiority; p = 0.001, t-test, 2 sided — p=.05 is the threshold for significance; Mean Difference (Final Values) = 7.78, 95% CI 2-sided [3.45 to 12.12]

ADVERSE EVENTS:
Time Frame: For any individual it was during the time of treatment and followup so 6 months.
Arm/Group | Experimental: 3RP Treatment | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 0/25 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/08/NCT02995408/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-14): https://cdn.clinicaltrials.gov/large-docs/08/NCT02995408/SAP_001.pdf
  • Informed Consent Form (2017-06-21): https://cdn.clinicaltrials.gov/large-docs/08/NCT02995408/ICF_002.pdf